CLINICAL TRIAL: NCT06134219
Title: A Mental Fatigue Course to Graves' Disease Patients With Mental Fatigue -a Randomized Controlled Study
Brief Title: Course for Brain Fatigue After Graves' Disease Controlled Study
Acronym: MF-Course
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MF-Course
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Graves Disease
Keywords: Mental fatigue
MeSH Terms: conditions — Graves Disease; Mental Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mental Fatigue course + Usual care in clinical care
  Interventions: Other: MF course; Other: Usual health care
- Control Group (Active Comparator): Usual care in clinical care
  Interventions: Other: Usual health care

INTERVENTIONS:
Other: MF course — A course consisting of six 2-hour-meetings every two-weeks with 10-15 participants (12 weeks in total). The meetings have different themes related to MF, such as understanding, practices for a deeper understanding of emotions, balance in everyday life with rest and activity, meditation practice to give time for brain rest, and mindfulness).
  Arms: Intervention
Other: Usual health care — The usual health care consists of one or few follow-up visits with blood tests at Sahlgrenska university hospital in Gothenburg or follow-up at the primary care after the end of treatment for Graves' treatment.

SUMMARY:
BACKGROUND. Mental fatigue (MF) is common in the most common form of hyperthyroidism, Graves' disease (GD). Clinically, MF is the primary mental symptom in patients with GD and is characterized by difficulties maintaining attention, exhaustion during cognitively demanding tasks, memory difficulties, irritability, and emotional lability. It may be the main contributing factor to the continued low quality of life in many patients with GD. MF can be measured with an MF score (MFS). The pathophysiology is unknown. There is no medical treatment, which requires patients to adapt to the situation.

AIM. In this project, the investigators want to test the hypothesis that mental fatigue improves - with secondary benefits on mental capacity, quality of life (QoL), and function - in patients with persistent mental fatigue in GD, through an MF course as an addition to standard care, compared to patients who receive only standard care. The investigators also test the hypothesis that the MF course is a cost-effective intervention.

METHOD. In a randomized controlled study, the investigators evaluate the effect of the MF course compared to standard care only in 96 patients with persistent MF in GD. Markers of mental health, QoL, and activity capacity are evaluated at baseline, 3, 6, and 12 months after intervention/inclusion. The primary outcome measure is MFS at 3 months.

CLINICAL SIGNIFICANCE. Patients report feeling neglected by healthcare for decades, and healthcare professionals are frustrated by the lack of guidance. Patient organizations highlight the need for research; they want mental symptoms to be characterized as a consequence of thyroid disease, they demand biomarkers, specific treatments, and personalized care. Our research group is working to address the cause of MF in GD and also to alleviate the symptoms. The MF course may prove to be an important tool that can be quickly implemented in clinical practice, especially in primary care. Our involvement in regional/national working groups will facilitate implementation in other units.

In this project, the investigators want to test the hypothesis that mental fatigue improves - with secondary benefits on mental capacity, quality of life (QoL), and function - in patients with persistent mental fatigue at GD, through an MF course as an addition to regular healthcare, compared to patients receiving only regular healthcare.

ELIGIBILITY:
Inclusion Criteria:

* 18-72 years old
* 15-72 months since first Graves' diagnosis
* high free thyroxin and thyroid antibodies (TRAb) at diagnosis
* euthyroid the last 6 months normal thyroid hormone levels at inclusion
* symptoms on MF in connection to Graves diagnosis
* MF-scale ≥10.5 points

Exclusion criteria:

* other diseases or situations that may be associated with mental fatigue (such as other active inflammatory disease, neurological disease)
* pregnancy
* lactation
* assessment that the patient cannot follow the study protocol.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Mental fatigue score | Change from baseline examined at 3 months follow-up.
  Scores at the Mental Fatigue Scale are compared between the intervention and the control group. Scores is between 0-42 and higher scores mean more brain fatigue.

SECONDARY OUTCOMES:
Comprehensive psychopathological rating questionnaire (CPRS) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS). Scores are compared between the intervention and the control group. Higher scores at the Comprehensive Psychopathological Rating Scale mean more symptoms of anxiety and depression. The Scores for anxiety is between 0-27 and for depression is between 0-27.
Comprehensive psychopathological rating questionnaire (CPRS) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS). Scores are compared between the intervention and the control group. Higher scores at the Comprehensive Psychopathological Rating Scale mean more symptoms of anxiety and depression. The Scores for anxiety is between 0-27 and for depression is between 0-27.
Comprehensive psychopathological rating questionnaire (CPRS) | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated questionnaire the Comprehensive Psychopathological Rating Scale (CPRS). Scores are compared between the intervention and the control group. Higher scores at the Comprehensive Psychopathological Rating Scale mean more symptoms of anxiety and depression. The Scores for anxiety is between 0-27 and for depression is between 0-27.
Coping Orientations to Problems Experienced (Brief cope) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire Brief cope. The Brief COPE is a shorter version of the COPE Inventory composed of 28-items rated on a 4-point ordinal scale that measure 14 subscales of coping style (2-items each). The overall mean is calculated with more than three being worse outcome. Coping strategies are compared between the intervention and the control group.
Coping Orientations to Problems Experienced (Brief cope) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire Brief cope. The Brief COPE is a shorter version of the COPE Inventory composed of 28-items rated on a 4-point ordinal scale that measure 14 subscales of coping style (2-items each).The overall mean is calculated with more than three being worse outcome. Coping strategies are compared between the intervention and the control group.
Coping Orientations to Problems Experienced (Brief cope) | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated questionnaire Brief cope. The Brief COPE is a shorter version of the COPE Inventory composed of 28-items rated on a 4-point ordinal scale that measure 14 subscales of coping style (2-items each).The overall mean is calculated with more than three being worse outcome. Coping strategies are compared between the intervention and the control group.
General Self-Efficacy Scale (GSE) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire General Self-Efficacy. Scores are compared between the intervention and the control group. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire General Self-Efficacy. Scores are compared between the intervention and the control group. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
General Self-Efficacy Scale (GSE) | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated questionnaire General Self-Efficacy. Scores are compared between the intervention and the control group. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Perceived Stress Scale (PSS-14) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14). Scores are compared between the intervention and the control group. The total score ranges between 0 and 56, with a higher score indicate more symptoms of stress.
Perceived Stress Scale (PSS-14) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14). Scores are compared between the intervention and the control group. The total score ranges between 0 and 56, with a higher score indicate more symptoms of stress.
Perceived Stress Scale (PSS-14) | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated questionnaire Perceived Stress Scale (PSS-14). Scores are compared between the intervention and the control group. The total score ranges between 0 and 56, with a higher score indicate more symptoms of stress.
Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39). Scores are compared between the intervention and the control group. ThyPRO scales is scored as a summary score and linearly transformed to range 0- 100. Higher scores at the Thyroid-specific Patient-Reported Outcome short-form means worse quality of life.
Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39). Scores are compared between the intervention and the control group. hyPRO scales is scored as a summary score and linearly transformed to range 0- 100. Higher scores at the Thyroid-specific Patient-Reported Outcome short-form means worse quality of life.
Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39) | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated questionnaire Thyroid-specific Patient-Reported Outcome short-form (ThyPro 39). Scores are compared between the intervention and the control group. hyPRO scales is scored as a summary score and linearly transformed to range 0- 100. Higher scores at the Thyroid-specific Patient-Reported Outcome short-form means worse quality of life.
Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). Scores are compared between the intervention and the control group. The range of each score is from 0 to 100, higher scores indicating better health.
Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). Scores are compared between the intervention and the control group. The range of each score is from 0 to 100, higher scores indicating better health.
Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated questionnaire the Graves' Ophthalmopathy Quality of Life Questionnaire (GO QoL). Scores are compared between the intervention and the control group. The range of each score is from 0 to 100, higher scores indicating better health.
EuroQol- health questionnaire (EQ-5D) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated questionnaire EuroQol- health (EQ-5D). Scores are compared between the intervention and the control group. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.
EuroQol- health questionnaire (EQ-5D) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated questionnaire EuroQol- health (EQ-5D). Scores are compared between the intervention and the control group. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.
EuroQol- health questionnaire (EQ-5D) | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated questionnaire EuroQol- health (EQ-5D). Scores are compared between the intervention and the control group. Each question may have 1 of 3-level answers, and a visual analog scale (VAS) on which patients can mark their current health state. The EQ-5D-3L index is calculated by subtracting the values of the descriptive EQ-5D system from the numerical value 1. This corresponds to the best possible health status, while an index value of <0 represents the worst possible health status.
Frenchay Activities Index (FAI) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated Frenchay Activities Index (FAI). Compare function and work ability between the intervention and the control group. Questionnaire consisting of 15 items on frequency of social everyday activities and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).
Frenchay Activities Index (FAI) | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated Frenchay Activities Index (FAI). Compare function and work ability between the intervention and the control group. Questionnaire consisting of 15 items on frequency of social everyday activities and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).
Frenchay Activities Index (FAI) | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated Frenchay Activities Index (FAI). Compare function and work ability between the intervention and the control group. Questionnaire consisting of 15 items on frequency of social everyday activities and the score is based on the frequency with which an activity has been performed during the previous 3 or 6 months. The total score ranges from 0 (inactive) to 45 (very active).
Work Productivity and Activity Impairment questionnaire (WPAI). Productivity and Activity Impairment questionnaire (WPAI) | Change from baseline examined at 3 months follow-up.
  Evaluated by the validated Work Productivity and Activity Impairment questionnaire (WPAI). Compare Work Productivity and Activity between the intervention and the control group.
  Four main outcomes can be generated from the WPAI-GH and expressed in percentages by multiplying the following scores by 100: 1) percent work time missed due to health = Q2/(Q2 + Q4) for those who were currently employed; 2) percent impairment while working due to health = Q5/10 for those who were currently employed and actually worked in the past seven days; 3) percent overall work impairment due to health Q2/(Q2 + Q4) + ((1 - Q2/(Q2 + Q4)) × (Q5/10)) for those who were currently employed; 4) percent activity impairment due to health Q6/10 for all respondents.
Evaluated by the validated Work Productivity and Activity Impairment questionnaire (WPAI). | Change from baseline examined at 6 months follow-up.
  Evaluated by the validated Work Productivity and Activity Impairment questionnaire (WPAI). Compare Work Productivity and Activity between the intervention and the control group.
  Four main outcomes can be generated from the WPAI-GH and expressed in percentages by multiplying the following scores by 100: 1) percent work time missed due to health = Q2/(Q2 + Q4) for those who were currently employed; 2) percent impairment while working due to health = Q5/10 for those who were currently employed and actually worked in the past seven days; 3) percent overall work impairment due to health Q2/(Q2 + Q4) + ((1 - Q2/(Q2 + Q4)) × (Q5/10)) for those who were currently employed; 4) percent activity impairment due to health Q6/10 for all respondents.
Work Productivity and Activity Impairment questionnaire (WPAI). Productivity and Activity Impairment questionnaire (WPAI) | Change from baseline examined at 12 months follow-up.
  Evaluated by the validated Work Productivity and Activity Impairment questionnaire (WPAI). Compare Work Productivity and Activity between the intervention and the control group.
  Four main outcomes can be generated from the WPAI-GH and expressed in percentages by multiplying the following scores by 100: 1) percent work time missed due to health = Q2/(Q2 + Q4) for those who were currently employed; 2) percent impairment while working due to health = Q5/10 for those who were currently employed and actually worked in the past seven days; 3) percent overall work impairment due to health Q2/(Q2 + Q4) + ((1 - Q2/(Q2 + Q4)) × (Q5/10)) for those who were currently employed; 4) percent activity impairment due to health Q6/10 for all respondents.
Days of sick-leave and cost related to health care and medication | Change from baseline examined at 3 months follow-up.
  Evaluated sick leave days between the intervention and the control group.
Days of sick-leave and cost related to health care and medication | Change from baseline examined at 6 months follow-up.
  Evaluated sick leave days between the intervention and the control group.
Days of sick-leave and cost related to health care and medication | Change from baseline examined at 12 months follow-up.
  Evaluated sick leave days between the intervention and the control group.
Levels of thyroid autoantibodies | Change from baseline examined at 3 months follow-up.
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid autoantibodies | Change from baseline examined at 6 months follow-up.
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid autoantibodies | Change from baseline examined at 12 months follow-up.
  Levels of thyroid autoantibodies, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid hormones | Change from baseline examined at 3 months follow-up.
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid hormones | Change from baseline examined at 6 months follow-up.
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Levels of thyroid hormones | Change from baseline examined at 12 months follow-up.
  Levels of thyroid hormones, analysed with the standard method of the laboratory at Sahlgrenska University Hospital, compared between the intervention and the control group.
Clinical Activity Score (CAS) | Change from baseline examined at 3 months follow-up.
  Comparison of Clinical Activity Score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-10 and higher scores mean more eye symptoms.
Clinical Activity Score (CAS) | Change from baseline examined at 6 months follow-up.
  Comparison of Clinical Activity Score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-10 and higher scores mean more eye symptoms.
Clinical Activity Score (CAS) | Change from baseline examined at 12 months follow-up.
  Comparison of Clinical Activity Score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-10 and higher scores mean more eye symptoms.
Severity score | Change from baseline examined at 3 months follow-up.
  Comparison of Severity score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-29 and higher scores mean more eye symptoms.
Severity score | Change from baseline examined at 6 months follow-up.
  Comparison of Severity score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-29 and higher scores mean more eye symptoms.
Severity score | Change from baseline examined at 12 months follow-up.
  Comparison of Severity score (a composite measure of ophthalmological signs and symptoms) between the intervention and the control group. Scores can be between 0-29 and higher scores mean more eye symptoms.
Mental fatigue score | Change from baseline examined at 6 months follow-up.
  Scores at the Mental Fatigue Scale are compared between the intervention and the control group. Scores can be between 0-42 and higher scores mean more brain fatigue.
Mental fatigue score | Change from baseline examined at 12 months follow-up.
  Scores at the Mental Fatigue Scale are compared between the intervention and the control group. Scores can be between 0-42 and higher scores mean more brain fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Filipsson Nyström, Principal Investigator — Sahlgrenska Universitet sjukhus
Locations (1):
- Agneta Lindo, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided